CLINICAL TRIAL: NCT05797233
Title: A Phase I Trial of Anti-CD19 and Anti-CD20 Bicistronic Chimeric Antigen Receptor T- Cells for Treating B-cell Malignancies
Brief Title: Trial of Anti-CD19 and Anti-CD20 Bicistronic Chimeric Antigen Receptor T Cells for Treating B-Cell Malignancies
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 10001524; 001524-C
Record Dates: First submitted 2023-04-01; First posted 2023-04-04 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01-09

CONDITIONS: Chronic Lymphocytic Leukemia; B-Cell Chronic Lymphocytic Leukemia; Lymphoma, B-Cell
Keywords: Immunotherapy; Autologous T Cells Infusion; Hu1928-Hu20BB; Adoptive T Cell Therapy; Gene Therapy
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1/Conditioning chemotherapy plus CAR T-cells dose escalation (Experimental): Escalating dose of anti-CD19 and anti-CD20 CAR T- cells/kg + conditioning chemotherapy
  Interventions: Biological: Anti-CD19 and anti-CD20 bicistronic CAR T- cells; Drug: Cyclophosphamide; Drug: Fludarabine
- 2/Conditioning chemotherapy plus CAR T-cells expansion phase (Experimental): MTD dose or Optimal dose of Anti-CD19 and anti-CD20 CAR T- cells/kg + conditioning chemotherapy
  Interventions: Biological: Anti-CD19 and anti-CD20 bicistronic CAR T- cells; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Biological: Anti-CD19 and anti-CD20 bicistronic CAR T- cells — 0.66x10^6 CAR+ T - 10x10^6 CAR+ T cells/kg (weight based dosing per cohort) infused on day 0
Drug: Cyclophosphamide — 500 mg/m^2 IV infusion over 30 minutes on days -5, -4 and -3
Drug: Fludarabine — 30 mg/m^2 IV infusion over 30 minutes administered immediately following the cyclophosphamide on days -5, -4,and -3

SUMMARY:
Background:

About 23,000 people die from B-cell cancers in the US each year. These cancers, often called leukemia or lymphoma, affect a type of white blood cell called B cells. These cancers are difficult to treat, and the therapies used can have bad side effects. Researchers want to try a new type of treatment. This new treatment uses a patient s own immune cells (T cells) that are modified to carry genes (chimeric antigen receptor, or CAR T cells) to kill cancer cells.

Objective:

To test a treatment using CAR T cells in people with B-cell cancers.

Eligibility:

People aged 18 to 75 years with a B-cell cancer that has not been controlled with standard therapies.

Design:

Participants will be screened. They will have:

Blood and urine tests.

A needle will be inserted to draw a sample of tissue from inside the hip bone.

For some patients, a needle will be inserted into their lower back to get a sample of the fluid around their spinal cord.

A tumor biopsy might be needed.

Imaging scans.

Tests of their heart function.

Participants will undergo apheresis: Blood will be drawn from a needle in an arm. The blood will pass through a machine that separates out the T cells. The remaining blood will be returned to the body through a second needle.

Participants will receive 2 chemotherapy drugs once a day for 3 days.

Participants will be admitted to the hospital for at least 9 days. Their T cells, now modified, will be infused back into their bloodstream through a tube placed in a large vein.

Follow-up visits will continue for 5 years, but patients will need to stay in touch with the CAR treatment team for 15 year.

DETAILED DESCRIPTION:
Background:

* Improved treatments for a variety of treatment-resistant malignancies including B-cell lymphomas, and chronic lymphocytic leukemia (CLL) are needed.
* A particular need is development of new treatments for chemotherapy-refractory B- cell malignancies.
* T- cells can be genetically modified to express chimeric antigen receptors (CARs) that specifically target malignancy-associated antigens.
* Autologous T- cells genetically modified to express CARs targeting the B-cell antigen CD19 have caused complete remissions in patients with leukemia or lymphoma. These results have established anti-CD19 CAR T- cells as an important therapy for relapsed lymphoma, but only about 40% of patients receiving anti-CD19 CAR T- cells have durable complete remissions.
* Most B-cell malignancies express CD19 and CD20, but expression of CD19 and CD20 can be lost or diminished.
* CD19 and CD20 are not expressed by normal cells except for B cells and some plasma cells.
* We have constructed a novel gene therapy construct that encodes a fully-human anti- CD19 CAR with a CD28 domain and a fully-human anti-CD20 CAR with a 4-1BB domain.
* T -cells expressing this CAR construct, called Hu1928-Hu20BB-Long, can specifically recognize CD19 and CD20-expressing target cells in vitro and eradicate CD19 or CD20-expressing tumors in mice.
* One CAR expressed in this CAR construct, Hu19-CD828Z has been tested in humans before. The other CAR in the total construct, Hu20-CD8BBZ-Long, has not been tested in humans before.
* Possible toxicities include cytokine-associated toxicities such as fever, hypotension, and neurological toxicities. Elimination of normal B cells is probable, and unknown toxicities are also possible.

Objective:

- Determine the safety of administering T-cells expressing a novel fully-human anti- CD19 and anti-CD20 CAR construct to participant with advanced B-cell malignancies.

Eligibility:

* Participant must have any B-cell lymphoma, or CLL/small lymphocytic lymphoma (SLL), or Gray-zone lymphoma. Lower grade lymphomas transformed to diffuse large B-cell lymphoma (DLBCL) are potentially eligible.
* Age >= 18 years of age and <=75 years of age at time of enrollment
* Participant must have malignancy that is measurable on a CT scan or by flow cytometry of bone marrow or blood.
* Participant must have a creatinine of 1.5 mg/dL or less and a normal cardiac ejection fraction.
* An ECOG performance status of 0-1 is required.
* No active infections are allowed including hepatitis B or hepatitis C.
* Absolute neutrophil count >=1000/microL, platelet count >=50,000/microL, hemoglobin >=8g/dL
* Serum ALT and AST less or equal to 3 times the upper limit of the institutional normal unless liver involvement by malignancy is demonstrated.
* At least 14 days must elapse between the time of any prior systemic treatment (including corticosteroids) and protocol-required leukapheresis or CAR T-cell infusion. In addition, sixty days must elapse from therapy with antibodies targeting CD19 or CD20 and CAR T-cell infusion, and at least 180 days must elapse since any prior CAR T-cell therapy or checkpoint therapy.
* The participant s malignancy will need to be assessed for CD19 and C20 expression by flow cytometry or immunohistochemistry performed at the NIH. If unstained, paraffin- embedded bone marrow or lymphoma tissue sections are available from prior biopsies, these can be used to determine CD19 and CD20 expression by immunohistochemistry; otherwise, Participant will need to come to the NIH for a biopsy to determine CD19 and CD20 expression. The sample for CD19 and CD20 expression must come from a biopsy obtained after any CD19 or CD20-targeted therapies such as monoclonal antibodies if such antibodies or CAR T-cell therapies have been received by the Participant.
* Either CD19 or CD20 expression must be uniform . Uniform CD19 or CD20 expression is defined as no obvious lymphoma population lacking antigen expression can be present.

Design:

* This is a phase I dose-escalation trial
* T-cells obtained by leukapheresis will be genetically modified to express the Hu1928- Hu20BB-Long CAR construct.
* Participants will receive a lymphocyte-depleting chemotherapy conditioning regimen with the intent of enhancing the activity of the infused CAR-expressing T- cells.
* The chemotherapy conditioning regimen is cyclophosphamide 500 mg/m^2 daily for 3 days and fludarabine 30 mg/m^2 daily for 3 days. Fludarabine will be given on the same days as the cyclophosphamide.
* Three days after the chemotherapy ends, participants will receive an infusion of anti- CAR- expressing T- cells .
* The initial dose level of this dose-escalation trial will be 0.66x10^6 CAR+ T- cells/kg of recipient bodyweight.
* The cell dose administered will be escalated until a maximum tolerated dose is determined.
* Following the T-cell infusion, there is a mandatory 9-day inpatient hospitalization to monitor for toxicity.
* Outpatient follow-up is planned for 2 weeks, and 1, 2, 3, 4, 6, 9, and 12 months after the CAR T-cell infusion; less frequent follow-up is required more than 1 year after infusion. Long-term gene-therapy follow-up for a total of 15 years after infusion is required.

ELIGIBILITY:
* INCLUSION CRITERIA:

Malignancy criteria

* CD19 and or CD20 expression is required. For all lymphoma types, eligibility criteria are met if there is uniform expression of both CD19 and CD20. Eligibility criteria are also met with expression of either CD19 or CD20. CD19 and/or CD20 expression must be "uniform". "Uniform" CD19 or CD20 expression is defined by CD19 and/or CD20 antigen expression on lymphoma cells with no obvious lymphoma population lacking antigen expression. Antigen expression can be assessed by either immunohistochemistry or flow cytometry.
* Pathology confirmed B-cell malignancy. Only when insufficient biopsy material is available to allow CD19 and CD20 expression assessment at the NIH, CD19 and/or CD20 staining performed at another institution can be used.
* At least 14 days must elapse between the time of any prior systemic treatment (including corticosteroids) and protocol-required leukapheresis or start of protocol conditioning chemotherapy.
* At least sixty days must elapse from therapy with antibodies targeting CD19 or CD20 and CAR T-cell infusion.
* At least 180 days must elapse after any prior CAR T-cell therapy, but otherwise, prior CAR T-cell therapy is allowed.
* Participants with DLBCL (including all subtypes such as primary mediastinal B-cell lymphoma and high-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangement) must have received at least two prior regimens at least one of which must have contained doxorubicin and an anti-CD20 monoclonal antibody.
* Follicular lymphoma participants must have received at least 2 prior regimens including at least 1 regimen with chemotherapy and 1 regimen with an anti-CD20 monoclonal antibody.
* Burkitt lymphoma participants must have had at least 1 prior cytotoxic chemotherapy- containing regimen that also contained an anti-CD20 monoclonal antibody.
* All participants with CLL or small lymphocytic lymphoma must have had at least 1 prior line of treatment, and these participants must have had progressive CLL/SLL after exposure to ibrutinib or another Bruton tyrosine kinase inhibitor and venetoclax.
* T-cell rich B-cell lymphoma is eligible if previously treated with at least 2 lines of therapy.
* Waldenstrom s macroglobulinemia/lymphoplasmacytic lymphoma patients are eligible if previously treated with at least 2 regimens including exposure to a monoclonal antibody, a bruton tyrosine kinase inhibitor, and cytotoxic chemotherapy.
* Participants with mantle cell lymphoma are eligible after receiving a Bruton tyrosine kinase (BTK) inhibitor, an anti-CD20 monoclonal antibody, and at least one of the following chemotherapy drugs: cytarabine, bendamustine, or an anthracycline.
* Other B-cell lymphoma types, including B-cell lymphoma unclassifiable with features intermediate between DLBCL and Hodgkin lymphoma (Gray zone), that are not specifically mentioned above are allowed if the participant has received at least 2 lines of therapy at least 1 of which must have contained cytotoxic chemotherapy.
* Primary central nervous system lymphoma patients are not eligible.

All participants must have measurable malignancy as defined by at least one of the criteria below.

- Lymphoma or leukemia masses that are measurable (minimum 1.5 cm in largest diameter) by CT scan is required for all diagnoses except CLL unless bone marrow or blood involvement with malignancy is detected. All masses must be less than or equal to

10.0 cm in the largest diameter.

* For a lymphoma mass to count as measurable malignancy, it must have abnormally increased metabolic activity when assessed by positron emission tomography (PET) scan. Exceptions to this rule are malignancies that do not consistently display increased metabolic activity on PET scans such as CLL/Small lymphocytic lymphoma.
* For CLL and lymphoma with only bone marrow and/or blood involvement no mass is necessary, but if a mass is not present, bone marrow and/or blood malignancy must be detectable by flow cytometry. Note that leukemia cells must make up 1% or less of peripheral blood lymphocytes within 2 weeks of the time of protocol enrollment in CLL participants for CLL participants to be eligible.

Other inclusion criteria:

* Greater than or equal to 18 years of age and less than or equal to 75 years of age.
* Clinical performance status of ECOG 0-1.
* Absolute neutrophil count greater than or equal to 1000/mm^3 without the support of filgrastim or other growth factors
* Platelet count greater than or equal to 50,000/mm^3 without transfusion support
* Hemoglobin greater than 8.0 g/dl
* Serum ALT and AST less or equal to 3 times the upper limit of the institutional normal unless liver involvement by malignancy is demonstrated. If liver involvement with malignancy is detected, ALT and AST must be less than or equal to 5 times the upper limit of normal.
* Serum creatinine less than or equal to 1.5 mg/dl
* Total bilirubin less than or equal to 2.0 mg/dl
* Room air oxygen saturation of 92% or greater
* Participants of child-bearing or child-fathering potential must be willing to practice birth control from the time of enrollment on this study and for four months after receiving the protocol treatment.
* A participant with a negative blood PCR test for hepatitis B DNA test can be enrolled. If hepatitis B DNA (PCR) testing is not available, participants with a negative hepatitis B surface antigen and negative hepatitis B core antibody can be enrolled.
* Participants must be tested for the presence of Hepatitis C antigen by PCR and be HCV RNA negative in order to be eligible. Only if Hepatitis C PCR testing is not available ina timely manner, participants who are Hepatitis C antibody-negative can be enrolled.
* Cardiac ejection fraction of greater than or equal to 50% by echocardiography and no evidence of hemodynamically significant pericardial effusion as determined by an echocardiogram within 4 weeks of treatment start.
* Participants must be able to understand and be willing to sign a written informed consent.
* Participants who have either been previously treated with genetically-modified T- cells including CAR T -cells of any specificity are potentially eligible if at least 180 days have elapsed since the prior infusion of genetically-modified T- cells. An exception to this is patients previously treated on this protocol can be re-treated on this protocol 8 weeks or more after the first treatment on this protocol.

EXCLUSION CRITERIA:

* Participants that require urgent therapy due to tumor mass effects or spinal cord compression.
* Participants must not have received any anti-CD20 or anti-CD19 antibody products in the past 60 days prior to CAR T-cell infusion.
* Participants that have active hemolytic anemia.
* HIV-positive patients.
* Participants with second malignancies in addition to their B-cell malignancy are not eligible if the second malignancy has required treatment (including maintenance therapy) within the past 3 years or is not in complete remission. There are two exceptions to this criterion: successfully treated non-metastatic basal cell or squamous cell skin carcinoma.
* Currently pregnant (confirmed with beta-HCG serum or urine pregnancy test performed at screening) or breastfeeding.
* Active uncontrolled systemic infections (defined as infections causing fevers within 48 hours of the date of planned protocol chemotherapy start and infections requiring intravenous antibiotics when intravenous antibiotics have been administered for less than 72 hours at the time of protocol chemotherapy start).
* Active coagulation disorders or other major uncontrolled medical illnesses of the cardiovascular, respiratory, endocrine, renal, gastrointestinal, genitourinary or immune system, history of myocardial infarction, history of ventricular tachycardia or ventricular fibrillation, active cardiac arrhythmias (active atrial fibrillation is not allowed, resolved atrial fibrillation not requiring current treatment is allowed (anticoagulants count as current treatment), active obstructive or restrictive pulmonary disease, active autoimmune diseases such as rheumatoid arthritis.
* Significant neurologic disorders that are not completely and permanently resolved and not requiring current treatment.
* Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
* Prior allogeneic stem cell transplant
* Systemic corticosteroid steroid therapy of any dose greater than 5 mg/day or more of prednisone or equivalent is not allowed within 14 days prior to the required leukapheresis, or the initiation of the conditioning chemotherapy regimen. Corticosteroid creams, ointments, and eye drops are allowed.
* Participants on systemic anticoagulant therapy except aspirin.
* History of severe immediate hypersensitivity reaction to any of the agents used in this study.
* Active central nervous system/brain metastases or cerebrospinal fluid malignancy.
* Checkpoint inhibitor drugs such as pembrolizumab or nivolumab or other antibodies targeting PD-1 or PDL-1 within 180 days of protocol enrollment. This is because of possible effects checkpoint inhibitor therapy could have on the patient s T- cells.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2023-08-28 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Determine the safety and feasibility of administering T cells expressing a novel fully-human anti-CD19 and anti-CD20 CAR construct to patients with advanced B-cell malignancies. | From time of lymphodepleting regimen through 30 days after the last CAR T infusion.
  Adverse Events (AE) by type and grade of toxicity

SECONDARY OUTCOMES:
Assess complete response rate | up to 5 years
  Complete Response rate (CR) in participants who receive subsequent infusion, up to 5 years after entry date for last participant
Assess overall response rate | up to 5 years
  Overall Response rate (ORR= CR + PR) will be recorded if ORR occurs at any response assessment time-point.
Assess duration of responses | up to 5 years
  Duration of response from date of response will be measured for no more than 5 years after the last participant has been enrolled on the trial.

CONTACTS AND LOCATIONS:
Overall Officials: James N Kochenderfer, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data will be available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_001524-C.html